CLINICAL TRIAL: NCT00901316
Title: Prevention of Recurrent Infections Caused by Community-Acquired Staphylococcus in Children 3 Months to 18 Years
Brief Title: Prevention of Recurrent Infections Caused by Community Acquired Staphylococcus Aureus (CA-SA) in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Sheldon Kaplan, Professor of Pediatrics, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Thrasher21631
Record Dates: First submitted 2009-05-11; First posted 2009-05-13 (Estimated); Results first posted 2016-11-07 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-09

CONDITIONS: Community-Acquired Staphylococcus Aureus
Keywords: Skin and Soft Tissue Infections; Abscesses; Boils; Clorox Baths; Colonization; Staph; MRSA; MSSA; Recurrent Infections; Prevention CA-SA Infections; Community-Acquired Staphylococcus in Children
MeSH Terms: conditions — Soft Tissue Infections; Abscess; Furunculosis; Staphylococcal Infections; Reinfection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Routine Measures (Experimental)
  Interventions: Procedure: Routine Measures Group
- Bleach Baths (Experimental)
  Interventions: Procedure: Bleach Bath Group (Bleach plus routine measures)

INTERVENTIONS:
Procedure: Routine Measures Group — Cultures will be obtained from the anterior nares of the nose, the throat and the groin using separate culturette swabs. S. aureus isolates will be identified and antibiotic susceptibility determined. Isolates will subsequently undergo testing for susceptibility to methicillin to determine if the isolate is an MSSA or MRSA strain. All patients and parents will be instructed orally and provided written instructions about routine measures employed for the prevention of S. aureus skin infections. Please see supplemental material from the publication Randomized Trial of "Bleach Baths" plus Routine Hygienic Measures vs Routine Hygienic Measures Alone for Prevention of Recurrent Infections Clinical Infectious Diseases 2014;58:679-682 for the details regarding routine measures.
  Other Names: Prevention of Infections Caused by CA-SA in Children.
  Arms: Routine Measures
Procedure: Bleach Bath Group (Bleach plus routine measures) — Cultures will be obtained from the anterior nares of the nose, the throat and the groin using culturette swabs. S. aureus isolates will be identified and antibiotic susceptibility determined. Isolates will subsequently undergo testing for susceptibility to methicillin to determine if the isolate is an MSSA or MRSA strain. Patients and parents will be instructed orally and provided written instructions about routine measures employed for the prevention of S. aureus skin infections. Patients will be given further oral and written instructions regarding clorox baths. Please see supplemental material from the publication Randomized Trial of "Bleach Baths" plus Routine Hygienic Measures vs Routine Hygienic Measures Alone for Prevention of Recurrent Infections Clinical Infectious Diseases 2014;58:679-682 for the details regarding instructions for bleach baths.
  Other Names: Clorox Baths
  Arms: Bleach Baths

SUMMARY:
The primary purpose of this study is to determine if adding bleach baths to routine ways for prevention of Staph infections is helpful. The amount added is a very weak amount. This would provide a relatively inexpensive method to help prevent recurrent skin infections caused by the Staph germ. The investigators will also be studying how often Staphylococcus aureus lives in the nose, throat, and groin area.

DETAILED DESCRIPTION:
In many areas of the United States, methicillin-resistant Staphylococcus aureus is now an established community pathogen (CA-MRSA). At Texas Children's Hospital (TCH), about 75% of S. aureus isolates recovered from healthy children with infections are CA-MRSA and > 90% of the CA-MRSA isolates are related to one clone, USA300, which also predominates throughout the U.S. From 8/05 to 7/06, 1400 children with CA-MRSA infection were seen at TCH; 60% were admitted to the hospital. Why the USA300 clone is so successful in spreading throughout the community is unclear, but it does harbor a unique set of genes not found in other S. aureus clones. The anterior nose in the most common area of the body colonized with S. aureus but it is not known if this is the primary site for colonization by CA-MRSA USA300 clone.

Approximately 3.5% of children at TCH have a proven recurrence of S. aureus infection within 12 months; we believe this is a minimal estimate and that overall at least 10% of children have recurrences. There is no consensus on the best strategies for preventing recurrent S. aureus infections or spread of S. aureus among family members. At TCH, in addition to routine preventative measures, we often recommend for the patients to take a bath at least twice a week in water to which one teaspoon of household bleach (Clorox) has been added per gallon of water. Anecdotally this approach has decreased the recurrence rate of S. aureus infections, but this common strategy among dermatologists has not been formally evaluated and is thus controversial.

Objectives

The primary objective is to test the hypothesis that in children who have a community-acquired Staphylococcus aureus (CA-SA) infection, sodium hypochlorite baths (Clorox) are a safe and effective component of a prevention strategy that will reduce recurrent medically attended skin and soft tissue infection (MA-SSI).

Specific Aims

1. Determine the recurrence rate (over a 12 month period) of medically attended skin and soft tissue infection visits in children initially evaluated in the TCH Emergency Center for whom a 3 month prevention strategy includes taking a bath twice a week in water to which sodium hypochlorite (Clorox) has been added and the recurrence rate in children for whom a similar prevention strategy has been recommended but without the bath component.
2. Determine the recurrence rate (over a 12 month period) of skin and soft tissue infection caused by CA-S. aureus in children for whom a 3-month prevention strategy includes taking a bath twice a week in water to which sodium hypochlorite (Clorox) has been added and the recurrence rate in children for whom a similar prevention strategy has been recommended but without the bath component.
3. Determine the + rates of S. aureus colonization of the anterior nares, pharynx, and groin for children being evaluated in the emergency center of Texas Children's Hospital (TCH) or admitted to TCH with suspected S. aureus infections.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy children 3 months to 18 years seen in the emergency center of Texas Children's Hospital with suspected CA-S. aureus infections
* Have a lesion which can be cultured (abscess or cellulitis with drainage, invasive infections)
* Can be evaluated and treated in the emergency center and be followed as outpatients
* Can be admitted to the hospital

Exclusion Criteria:

* Children less than 3 months old or greater than 18 years
* Immune deficiency or underlying condition other than reactive airway disease or simple eczema which is not being followed by a dermatologist
* Patient has a history of 2 or more previous skin or soft tissue infections
* Children with one previous episode whose family may have already employed the sodium hypochlorite baths
* Families without a bathtub or running water
* Families without a phone or primary care physician
* Families unable or unwilling to comply with the prevention measures
* Hypersensitivity to sodium hypochlorite

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 987 (Actual)
Dates: Start 2009-06; Primary Completion 2012-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon L Kaplan, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Baylor College of Medicine, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- See also: NCT00179959 — http://www.clinicaltrials.gov

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children with probable community-associated Staphylococcus aureus skin and soft tissue or invasive infections were randomized to routine daily hygienic measures with or without "bleach baths" twice a week for 3 months.
Groups:
- Routine Measures: Routine Measures Group: Cultures will be obtained from the anterior nares of the nose, the throat and the groin using separate culturette swabs. S. aureus isolates will be identified and antibiotic susceptibility determined. Isolates will subsequently undergo testing for susceptibility to methicillin to determine if the isolate is an MSSA or MRSA strain. All patients and parents will be instructed orally and provided written instructions about routine measures employed for the prevention of S. aureus skin infections.
- Bleach Baths: Bleach Bath Group: Cultures will be obtained from the anterior nares of the nose, the throat and the groin using culturette swabs. S. aureus isolates will be identified and antibiotic susceptibility determined. Isolates will subsequently undergo testing for susceptibility to methicillin to determine if the isolate is an MSSA or MRSA strain. Patients and parents will be instructed orally and provided written instructions about routine measures employed for the prevention of S. aureus skin infections. Patients will be given further oral and written instructions regarding clorox baths.
Period: Overall Study
Arm/Group | Routine Measures | Bleach Baths
Started | 492 | 495
Completed | 492 | 495
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: We needed to enroll 482 children in each arm to detect a 50% reduction in recurrences with 90% power, assuming a 12-month recurrence rate of 14% in the hygiene only group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Routine Measures | Bleach Baths | Total
Number analyzed (Participants) | 492 | 495 | 987
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 492 | 495 | 987
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 1.92 [.26 to 18.8] | 1.8 [.27 to 17.9] | 1.85 [.26 to 18.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 253 | 276 | 529
  Male | 239 | 219 | 458
Region of Enrollment [Number; unit: participants]
  United States | 492 | 495 | 987

OUTCOME MEASURES:

1. Primary Outcome: Medically Attended Skin and Soft Tissue Infections (MA-SSI)
Description: Medically attended skin and soft tissue infections (MA-SSI) which is defined as a skin or soft tissue infection that has been evaluated and treated by a medical professional in an office, clinic, urgent care or emergency center setting.
Time Frame: From time of enrollment until the first MA-SSI or 12 months following enrollment, whichever came first.
Measure: Number (95% Confidence Interval); unit: percentage of partipants
Arm/Group | Routine Measures | Bleach Baths
Number analyzed (Participants) | 492 | 495
percentage of partipants | 20.9 [17.3 to 24.5] | 17 [13.7 to 20.3]

ADVERSE EVENTS:
Arm/Group | Routine Measures | Bleach Baths
Serious Adverse Events (participants affected / at risk) | 0/492 | 0/495
Other Adverse Events (participants affected / at risk) | 0/492 | 1/495
OTHER ADVERSE EVENTS (reported when occurring in more than .01% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Routine Measures (N=492) | Bleach Baths (N=495)
Burning eyes (Eye disorders) | 0 | 1 — Burning eyes

LIMITATIONS AND CAVEATS:
We were limited in detecting decreases in recurrent MA-SSTI < 50% because of the large sample size required.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No